CLINICAL TRIAL: NCT01253564
Title: An Open-label, Pilot Study of RO5185426 in Previously Treated Metastatic Melanoma Patients With Brain Metastases
Brief Title: A Study of RO5185426 in Previously Treated Melanoma Patients With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO25653
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO5185426

INTERVENTIONS:
Drug: RO5185426 — 960 mg b.i.d. orally

SUMMARY:
This open-label study will assess the safety and efficacy of RO5185426 in previously treated metastatic melanoma patients with brain metastases. Patients will receive RO5185426 at a dose of 960 mg twice daily orally until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Metastatic melanoma (Stage IV, American Joint Committee on Cancer) with BRAF mutation (cobas 4800 BRAF V600 Mutation Test)
* Brain metastases for which surgical resection is not a treatment option
* Patients must have failed at least one previous treatment for brain metastases
* Requiring corticosteroids for symptom control
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Increasing corticosteroid dose during the 7 days prior to study entry
* Previous malignancy within the past 2 years, except for basal or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix
* Concurrent administration of any anticancer therapies other than those administered in the study
* Clinically significant cardiovascular disease or event within the 6 months prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2012-03-14 (Actual); Study Completion 2012-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Switzerland (2):
  - CHUV; Departement d'Oncologie, Lausanne
  - Universitätsspital Zürich; Dermatologische Klinik, Zurich

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib: Participants received vemurafenib tablets, 960 milligrams (mg), twice daily (BID), orally continuously until disease progression, unacceptable toxicity, withdrawal of consent, death, other reason deemed by investigator or study termination by the Sponsor.
Period: Overall Study
Arm/Group | Vemurafenib
Started | 24
Completed | 0
Not Completed | 24
Not completed — Disease Progression | 22
Not completed — Withdrawal by Subject | 1
Not completed — Serious Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received at least one dose of study medication.
Groups:
- Vemurafenib: Participants received vemurafenib tablets, 960 mg, BID, orally continuously until disease progression, unacceptable toxicity, withdrawal of consent, death, other reason deemed by investigator or study termination by the Sponsor.
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: AE:any unfavorable and unintended sign, symptom, or disease associated with use of study drug, regardless of relation to study drug. Pre-existing conditions that worsened and laboratory or clinical tests that resulted in change in treatment or discontinuation from study drug were reported as AEs. Serious AE: resulted in death, life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect or was medically significant. Grade-1:discomfort but no disruption of normal daily activity. Grade-2:discomfort sufficient to reduce or affect daily activity,no intervention indicated.Grade-3:inability to perform normal daily activity,intervention indicated.Grade-4:immediate threat to life or leading to permanent mental or physical condition that prevented performing normal daily activities.Grade 5: death. Any AE included participants with serious and non-serious AE.
Time Frame: From baseline up to last dose (0.1 to 11.3 months) plus 28 days
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants
  Any AEs | 96
  Drug-related AEs | 83
  AEs of Grade 1 and 2 | 92
  AEs of Grade 3 | 17
  AEs of Grade 5 | 4
  SAEs | 58
  Drug-related SAEs | 17
  AEs that led to Study Drug Discontinuation | 4
  AEs that led to Study Drug Reduction | 0
  AEs that led to Study Drug Interruption | 4

2. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) by Disease Site
Description: Objective response was assessed by the investigator according to Response Evaluation Criteria in Solid Tumours (RECIST) (Version 1.1). CR was defined as disappearance of all target and non-target lesions and no new lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Best overall response was calculated separately for brain, other sites (extracranial) and whole body. Percentage of participants with 95 percent (%) Clopper-Pearson confidence interval (CI) are reported.
Time Frame: Baseline, Week 4, Week 8 and thereafter every 8th week until progressive disease, unacceptable toxicity, consent withdrawal, death or other reasons deemed by the investigator (up to 16 months)
Population: Safety population. Here, 'n' signifies the number of participants with measurable disease at baseline for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants
  Brain (n=19) | 15.8 [3.4 to 39.6]
  Extracranial (n=21) | 61.9 [38.4 to 81.9]
  Whole body (n=24) | 41.7 [22.1 to 63.4]

3. Secondary Outcome: Duration of Response by Disease Site
Description: Duration of response was defined as the time interval between the date of the earliest qualifying response and the date of progressive disease (PD) or death, only for those participants whose best overall response was CR or PR. CR and PR were assessed by investigator according to RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. PD was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 millimeter (mm), progression of existing non-target lesions, or presence of new lesions. Duration of response was calculated by Kaplan-Meier estimates separately for brain, other sites (extracranial) and whole body.
Time Frame: Baseline, Week 4, Week 8 and thereafter every 8th week until progressive disease or death (up to 16 months)
Population: Safety population. Here, 'n' signifies number of participants with best overall response of CR or PR for specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
months
  Brain (n=3) | 4.4 [2.1 to 4.6]
  Extracranial (n=13) | 3.8 [2.7 to 5.3]
  Whole body (n=10) | 3.7 [2.7 to 4.8]

4. Secondary Outcome: Time to Response by Disease Site
Description: Time to response was defined as the interval between the date of first treatment and the date of first documentation of CR or PR (whichever occurred first). CR and PR were assessed by investigator according to RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Time of response was calculated by Kaplan-Meier estimates separately for brain, other sites (extracranial) and whole body.
Time Frame: as for outcome 2
Population: Safety population. Here, 'n' signifies number of participants with measurable disease for specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
months
  Brain (n=19) | NA [NA to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  Extracranial (n=20) | 1.4 [0.9 to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  Whole body (n=23) | 5.5 [1.8 to NA] — Estimate not available due to insufficient follow-up to allow estimation.

5. Secondary Outcome: Duration of Stable Disease (SD) by Disease Site
Description: Duration of SD was defined as the time between the first documented date of SD and date of PD or death from any cause. SD was defined (according to RECIST version 1.1) as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. PD was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. Duration of SD was calculated by Kaplan-Meier estimates separately for brain, other sites (extracranial) and whole body.
Time Frame: as for outcome 2
Population: Safety Population. Here, 'n' signifies number of participants with measurable disease at baseline for specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
months
  Brain (n=13) | 5.5 [4.1 to 5.6]
  Extracranial (n=6) | 3.9 [2.3 to 12.1]
  Whole body (n=9) | 3.9 [3.7 to 5.6]

6. Secondary Outcome: Time to New Lesion by Disease Site
Description: Time to new lesions was defined as the interval between the date of first treatment and the date of first documentation of new lesions. Time to new lesion was calculated by Kaplan-Meier estimates separately for brain, other sites (extracranial) and whole body.
Time Frame: Baseline, Week 4, Week 8 and thereafter every eighth week until progressive disease, unacceptable toxicity, consent withdrawal, death or other reasons deemed by the investigator (up to 16 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
months
  Brain (n=23) | 5.6 [3.9 to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  Extracranial (n=23) | NA [NA to NA] — Estimate not available due to insufficient follow-up to allow estimation.
  Whole body (n=23) | 5.6 [3.9 to NA] — Estimate not available due to insufficient follow-up to allow estimation.

7. Secondary Outcome: Percentage of Participants With Disease Progression or Death by Disease Site
Description: Disease progression (according to RECIST version 1.1) was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study or absolute increase and at least 5 mm, progression of existing non-target lesions, or presence of new lesions. Percentage of participants with disease progression by brain, other sites (extracranial) and whole body are reported.
Time Frame: as for outcome 2
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants
  Brain | 100
  Extracranial | 83.3
  Whole body | 100

8. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval between the date of the first treatment and the date of progression or death from any cause, whichever occurred first. Disease progression (according to RECIST version 1.1) was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study or absolute increase and at least 5 mm, progression of existing non-target lesions, or presence of new lesions. PFS was calculated by Kaplan-Meier estimates separately for brain, other sites (extracranial) and whole body.
Time Frame: as for outcome 6
Population: Safety Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
months
  Brain | 4.3 [3.1 to 5.5]
  Extracranial | 4.6 [3.1 to 5.6]
  Whole body | 3.9 [3.0 to 5.5]

9. Secondary Outcome: Percentage of Participants Who Died
Description: Percentage of participants who died due to any reason are reported.
Time Frame: Baseline up to end of the study and every 3 months during follow-up (up to 16 months)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants | 79.2

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first treatment to the date of death, regardless of the cause of death. Participants who discontinued the study treatment for any reason other than withdrawal of consent were continued to be followed for survival. The end of study occurred when all participants had been followed for a period of 6 months, had died, withdrawn consent or were lost to follow-up, whichever occurred first. OS was calculated by Kaplan-Meier estimates.
Time Frame: From start of treatment up to end of the study and every 3 months during follow up (up to 16 months)
Population: Safety population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
months | 5.3 [3.9 to 6.6]

11. Secondary Outcome: Percentage of Participants With Improvement in Total Daily Dose of Corticosteroids
Description: An improvement in corticosteroid dose was defined as a dose reduction of at least 33% of baseline dose for at least 28 days or stopping use completely. Percentage of participants and 95% Clopper-Pearson CI are reported.
Time Frame: Baseline, every week during the first 8 weeks and every second week thereafter up to last dose (0.1 to 11.3 months) plus 28 days
Population: Safety Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants | 66.7 [44.7 to 84.4]

12. Secondary Outcome: Percentage of Participants With Improvement in Total Daily Dose of Narcotic Pain Analgesic
Description: An improvement in narcotic pain analgesics was defined as a dose reduction of at least 33% of baseline dose for at least 28 days or stopping use completely.
Time Frame: as for outcome 11
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants | 8.3

13. Secondary Outcome: Percentage of Participants With Improvement in Visual Analog Scale (VAS) Assessment of Pain
Description: VAS is a measure of pain intensity. The participant was asked to mark on a 100 mm line where their pain level was on the day they completed the scale. The beginning of the line represented no pain and the end of the line represented maximum pain. Total score ranged from 0 - 100. Reported values are decrease in VAS of greater than (>) 20 mm or >30 mm from baseline.
Time Frame: Baseline; Day 1 of Cycles 2-8 (28-day cycle) and at the end of study visit (up to 16 months)
Population: Safety population. Here, 'n' signifies number of participants with available data for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants
  Decrease of > 20 mm: Any visit (n=24) | 25.0
  Decrease of >30 mm: Any visit (n=24) | 20.8
  Decrease of > 20 mm: Cycle 2 - Day 29 (n=23) | 26.1
  Decrease of >30 mm: Cycle 2 - Day 29 (n=23) | 13.0
  Decrease of > 20 mm: Cycle 3 - Day 57 (n=20) | 20.0
  Decrease of >30 mm: Cycle 3 - Day 57 (n=20) | 20.0
  Decrease of > 20 mm: Cycle 4 - Day 85 (n=18) | 16.7
  Decrease of >30 mm: Cycle 4 - Day 85 (n=18) | 16.7
  Decrease of > 20 mm: Cycle 5 - Day 113 (n=13) | 7.7
  Decrease of >30 mm: Cycle 5 - Day 113 (n=13) | 7.7
  Decrease of > 20 mm: Cycle 6 - Day 141 (n=10) | 10.0
  Decrease of > 30 mm: Cycle 6 - Day 141 (n=10) | 10.0
  Decrease of > 20 mm: Cycle 7 - Day 169 (n=8) | 12.5
  Decrease of > 30 mm: Cycle 7 - Day 169 (n=8) | 0.0
  Decrease of > 20 mm: Cycle 8 - Day 197 (n=4) | 25.0
  Decrease of >30 mm: Cycle 8 - Day 197 (n=4) | 25.0
  Decrease of > 20 mm: End of Study (n=12) | 16.7
  Decrease of >30 mm: End of Study (n=12) | 16.7

14. Secondary Outcome: Percentage of Participants With Improvement in Physician's Assessment of Global Performance Status
Description: Physician's Assessment of Global Performance Status was assessed on 7 point scale (1- Very much better, 2-Much better, 3-A little better, 4-No change, 5-A little worse, 6-Much worse, 7- Very much worse). An improvement was classed as a difference from baseline of at least -1 point. Percentage of participants with 95% Clopper-Pearson CI were reported for participants with improvement in Physician's Assessment of Global Performance Status at any visit.
Time Frame: Baseline, Day 1 of every 28-day cycle, at end of study and at the 28-day follow-up visit (up to 16 months)
Population: Safety population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 24
percentage of participants | 83.3 [58.6 to 96.4]

ADVERSE EVENTS:
Time Frame: From baseline up to last dose (0.1 to 11.3 months) plus 28 days
Arm/Group | Vemurafenib
Serious Adverse Events (participants affected / at risk) | 14/24
Other Adverse Events (participants affected / at risk) | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=24)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Epilepsy (Nervous system disorders) | 5
Cerebral disorder (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Erysipelas (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Confusional state (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=24)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 5
Solar dermatitis (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Dizziness (Nervous system disorders) | 5
Epilepsy (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Ageusia (Nervous system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Oral candidiasis (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Fatigue (General disorders) | 4
Oedema peripheral (General disorders) | 4
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Sleep disorder (Psychiatric disorders) | 3
Haematoma (Vascular disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 2
Alanine aminotransferase increased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.